CLINICAL TRIAL: NCT05343494
Title: Maternal Health Diabetes Prevention Project Pilot Study
Brief Title: Maternal Health Diabetes Prevention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: Westat (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021-1234; OT2HL158287 (NIH)
Record Dates: First submitted 2022-04-04; First posted 2022-04-25 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-04

CONDITIONS: Gestational Diabetes; PreDiabetes; Hyperglycemia; Glucose Intolerance During Pregnancy
Keywords: Diabetes Prevention Program; Behavioral Intervention; Diet; Physical Activity; Special Supplemental Nutrition Program for Women, Infants, and Children (WIC)
MeSH Terms: conditions — Diabetes, Gestational; Prediabetic State; Hyperglycemia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle Intervention (Experimental): The intervention has been modified from a subset of sessions from the National DPP Prevent T2 Curriculum (an adapted DPP for community settings that improves cardiometabolic outcomes and is implemented nationwide).
  The intervention will consist of 8 weekly sessions. The first session will be one-on-one and subsequent sessions will be in small groups. Sessions 1, 2, and 6 will be in-person and other sessions will be held by Zoom.
  Interventions: Behavioral: Lifestyle Intervention

INTERVENTIONS:
Behavioral: Lifestyle Intervention — The intervention has been modified from a subset of sessions from the National DPP Prevent T2 Curriculum (an adapted DPP for community settings that improves cardiometabolic outcomes and is implemented nationwide).
  The intervention will consist of 8 weekly sessions. The first session will be one-on-one and subsequent sessions will be in small groups. Sessions 1, 2, and 6 will be in-person and other sessions will be held by Zoom.

SUMMARY:
The aim of this project is to use the Exploration, Preparation, Implementation, Sustainment (EPIS) framework to collect pilot data on the implementation of a Diabetes Prevention Program-like intervention in the Women, Infants, and Children (WIC) program.

DETAILED DESCRIPTION:
In this study, investigators will pilot a 2-month Diabetes Prevention Program-like program (delivered by WIC staff) to 20 women with recent gestational diabetes (6 weeks to 12 months postpartum) who receive WIC services.

The goal of this pilot is to evaluate the feasibility, acceptability, appropriateness, fidelity of implementing this intervention in the setting of WIC clinics and feasibility of conducting a larger-scale study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* 6 weeks to 12 months postpartum
* Medical record documented diagnosis of GDM during most recent pregnancy
* Access to a device that can access the internet
* English speaking

Exclusion Criteria:

* Pregnant or planning to become pregnant in the next two months
* Planning to move out of the area in the next two months
* Self-report of diagnosed diabetes
* Use of glucose-lowering medications
* Plasma glucose >200 mg/dL and classic symptoms of hyperglycemia (thirst, polyuria, weight loss, blurry vision) or HbA1c >6.5% (based on screening visit blood draw)
* Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Fidelity - sessions attended | 8-week intervention
  Number of sessions attended throughout the 8 week intervention

SECONDARY OUTCOMES:
Fidelity - sessions held | 8-week intervention
  Number of sessions held throughout the 8 week intervention
Fidelity - session content | 8-week intervention
  Assessment of whether key concepts were covered during sessions
Intervention feasibility | 2-month data collection visit
  Feasibility questionnaire delivered to participants and staff delivering the intervention
Intervention appropriateness | 2-month data collection visit
  Appropriateness questionnaire delivered to participants and staff delivering the intervention
Intervention acceptability | 2-month data collection visit
  Acceptability questionnaire delivered to participants and staff delivering the intervention

OTHER OUTCOMES:
Diet | 2 months
  2-month change in self-reported dietary intake assessed by Dietary Screener Questionnaire
Physical activity | 2 months
  2-month change in self-reported physical activity (metabolic equivalents) assessed by International Physical Activity Questionnaire
Weight | 2 months
  Change in weight from baseline to 2-month visit
Hemoglobin A1c | 2 months
  Change in hemoglobin A1c from baseline to 2-month visit
Fasting plasma glucose | 2 months
  Change in fasting plasma glucose from baseline to 2-month visit
Recruitment yield | Pre-enrollment (before enrollment into the study)
  Yield of participants recruited (out of number of prescreening calls, screening visits)
Retention | Through 2-month study period
  Proportion of participants retained to end of 2-month study
Staff time involved in intervention delivery | Through 2-month study period
Staff time involved in recruitment | Pre-enrollment (before enrollment into the study)
Staff time involved in data collection | Through 2-month study period
Qualitative interviews | 2 months
  Qualitative interviews with staff delivering intervention and WIC participants participating in the intervention. Topics covered: barriers and facilitators, intervention feasibility, appropriateness and acceptability, fidelity, potential for scalability and sustainability, usability of the technology and apps used in the intervention, recommendations to improve the intervention/implementation,

CONTACTS AND LOCATIONS:
Locations (1):
- Tulane Office of Health Research, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No